CLINICAL TRIAL: NCT03764956
Title: Comparison of Efficacy of Low Glycemic Index Therapy and Modified Atkins Diet Among Children With Drug Resistant Epilepsy: A Randomized Non-inferiority Trial
Brief Title: Comparison of Efficacy of LGIT and MAD Among Children With Drug Resistant Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, Chief, Child Neurology Division, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECPG/504/10/2018
Record Dates: First submitted 2018-11-04; First posted 2018-12-05 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Drug Resistant Epilepsy; Ketogenic Dieting
Keywords: MAD; LGIT
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Open label randomized non inferiority trial with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Index therapy (Experimental): Specific dietary therapy called Low glycemic Index Therapy (LGIT) which provides diet including food items with glycemic index less than 50 only
  Interventions: Other: Low glycemic Index Therapy (LGIT)
- Modified Atkins Diet (Active Comparator): Specific dietary therapy called Modified Atkins Diet (MAD) which provides diet with restricted carbohydrates upto 20 grams per day and increased fat and protein ratio
  Interventions: Other: Modified Atkins Diet (MAD)

INTERVENTIONS:
Other: Low glycemic Index Therapy (LGIT) — Specific dietary therapy called Low glycemic Index Therapy (LGIT) which provides diet including food items with glycemic index less than 50 only. For this purpose, various dietary menus will be provided to the parents.
  Arms: Low Glycemic Index therapy
Other: Modified Atkins Diet (MAD) — Specific dietary therapy called Modified Atkins Diet (MAD) which provides diet with restricted carbohydrates upto 20 grams per day and increased fat and protein ratio. For this purpose, various dietary menus will be provided to the parents.
  Arms: Modified Atkins Diet

SUMMARY:
To compare the efficacy of two less restrictive dietary therapies - LGIT and MAD, used for treatment of drug resistant epilepsy in children

DETAILED DESCRIPTION:
Up to one third of patients with epilepsy progress to drug resistant epilepsy (DRE). Current treatment options for DRE include epileptic surgery and dietary therapy. Classic KD (Ketogenic diet) is the most studied dietary therapy but the stringent restrictions and practical difficulty makes it difficult to follow. So less restrictive diets like MAD and LGIT were introduced. These are reported to have less adverse effects also. But no published study has ever been conducted comparing these two diets head to head.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-15 years with drug resistant epilepsy
* Willing to come for regular follow-up according to study protocol Drug resistant epilepsy defined as
* Seizure frequency >4 seizures per month, while on optimal doses of at least 2 prescribed antiepileptic drugs
* For West syndrome, drug resistant epilepsy will be defined as more than 4 clusters of spasms per month despite treatment with antiepileptic drugs and either ACTH(Adrenocorticotrophic hormone) or Vigabatrin

Exclusion Criteria:

* Surgically remediable causes for DRE
* Inborn errors of metabolism
* Previously received KD, MAD or LGIT
* Known case of

  1. Chronic kidney disease
  2. Chronic liver disease/GI illness
  3. Congenital/acquired heart disease
  4. Chronic respiratory illness

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of seizure reduction from baseline at 24 weeks of therapy | At the end of 24 weeks of dietary therapy
  Mean weekly seizure reduction at 24 weeks divided by Mean weekly seizure measured at baseline multiplied by 100

SECONDARY OUTCOMES:
Proportion of children who achieve >50% seizure reduction | At the end of 24 weeks of dietary therapy
  Number of children with >50% reduction divided by number of children in each arm
Incidence of adverse events | At the end of 24 weeks of dietary therapy
  Routine hemogram, Renal function test (RFT), Liver function test (LFT) and lipid profile will be assessed for any alterations. Adverse events, vomiting, constipation and diarrhea will be checked by parents record
Compliance of participants with dietary therapy in each arm will be determined each week, whether satisfactory or unsatisfactory | At the end of 24 weeks of dietary therapy
  Weekly compliance assessment of each participant will be done
Change in Social quotient(SQ) with each dietary therapies | At the end of 24 weeks of dietary therapy
  Proportion of children with improvement in Social quotient (SQ) assessed by Vineland Social Maturity Scale (VSMS) at 24 weeks. VSMS consists of 8 subsets - Communication skills, General self-help ability, Locomotion skills, Occupation skills, Self-direction, Self-help eating, Self-help dressing, Socialization skills. Social age is calculated by adding the scores of all subsets. Social quotient (SQ) is calculated by social age divided by chronological age multiplied by 100.
Change in Quality of Life of participants who are less than 4 years of age at 24 weeks as compared to baseline | At the end of 24 weeks of dietary therapy
  In children less than 4 years quality of life is assessed by PedsQL (Pediatric Quality of life inventory). PedsQL consists of 21 questions each having 5 responses with scores 0,1,2,3 and 4. Minimum score is 0 and maximum is 84. Quality of life is poor with larger score.
Change in Quality of Life of participants who are more than or equal to 4 years of age at 24 weeks as compared to baseline | At the end of 24 weeks of dietary therapy
  In children with age 4 years or more, QOLCE 55 (Quality of life in childhood epilepsy questionnaire) is used to assess quality of life. QOLCE 55 consists of 55 questions which are classified into 4 categories. Each question have 5 responses with scores as 0,25,50,75 and 100. Mean score of each category is calculated and final score calculated by mean of the scores of 4 categories. Minimum score is 0 and maximum is 100. Quality of life is better with larger score.
Change in Quality of Life of caregivers at 24 weeks as compared to baseline | At the end of 24 weeks of dietary therapy
  Quality of life of caregivers is assessed by WHOQOL-BREF. WHOQOL BREF contains 26 items categorized into 4 domains. For each question response is scored 1,2,3,4 or 5. Total raw score is then calculated and is converted to transformed score. Minimum score is 0 and maximum is 100. Quality of life is poor with smaller score.
Gut microbiota (GM) analysis pre and post dietary therapy | At the end of 24 weeks of dietary therapy
  Changes in percentage distribution of various micro organisms in gut microbiota after dietary therapy as compared to baseline GM
Change in behavioral abnormalities with each dietary therapy | At the end of 24 weeks of dietary therapy
  Behavior assessment is done using Child behavior check list (CBCL).This questionnaire contains 100 and 113 questions for age groups of 1 ½ - 5 years and 6-18 years respectively. Score of 2 will be given for a response of 'very true', 1 for a response of 'somewhat true' and 0 for 'not true'. Total score is obtained by adding all the subsets. Subsets for age 1.5 years to 5 years include - Emotionally reactive, anxious/depressed, somatic complaints, withdrawn, sleep problems, attention problems, aggressive behavior and other problems. Subsets for age 6 years to 12 years include - Anxious/Depressed, withdrawn, somatic complaints, social problems, thought problems, attention problems, rule breaking behavior, aggressive behavior, other problems. Raw score is then converted to T score according to the published charts. Minimum T score is 28 and maximum is 100. Larger score indicates more behavioral problems.

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - AIIMS, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Undecided